CLINICAL TRIAL: NCT03874975
Title: Combined Oral Vitamin D and UVB Versus Alone in Treatment of Psoroasis Vulgaris
Brief Title: Combined Oral Vitamin D and UVB Versus UVB Alone in Treatment of Psoriasis Vulgaris
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Meryhan Ashraf Abdelazeem, principal Investigator, Assiut University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: vit D and UVB in psoriasis
Record Dates: First submitted 2019-03-06; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: 40 patients divided into two groups : group 1 :20 patients underoral vitamin D and UVB group 2 : 20 patients under uvb alone in psoriatic patients
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: oral vitamin D — vitamin D and UVB versus UVB alone in psoriatic patients and evaluate patients by PASI score before and after treatment and measure serum vitamin D before and after treatment
  Other Names: narrow band UVB

SUMMARY:
To compare the results of vitamin D plus UVB in treatment of psoriasis vulgaris with the results of UVB alone to study the relation between serum vitamin D and PASI score before and after treatment.

DETAILED DESCRIPTION:
Psoriasis is a chronic immune-mediated inflammatory skin disease, with a prevalence of about 2%-3% in the general population. The primary manifestation of psoriasis most commonly manifests on the skin, although inflammatory processes can occur also in other organs .

Vitamin D, also known as the sunshine vitamin, has long been known to be a hormone that regulates calcium-phosphorous homeostasis and safeguards the integrity of the skeletal system . The epidermis is the natural source of vitamin D synthesis by the action of ultraviolet light (UV) B of the sun or other UVB source . On the other hand, evidence is accumulating that vitamin D might represent a key modulator of immune and inflammation mechanisms . Recently, a role for vitamin D in the pathogenesis of different skin diseases, including psoriasis, has been reported.

Psoriasis lesions are characterized by hyper-proliferation with incomplete differentiation of epidermal keratinocytes and decreased keratinocyte apoptosis, associated with inflammatory cellular infiltrate in both dermis and epidermis . Psoriasis Area and Severity Index (PASI) score is currently the preferred method for the assessment of the disease severity and extent .

Physiologically, the active form of vitamin D and its receptor regulate the differentiation and proliferation of keratinocytes, the balance of the cutaneous immune system and the process of apoptosis.

Several studies identified an association between polymorphisms of vitamin D receptor (VDR) and psoriasis susceptibility .The 1,25(OH)D has been shown to exert anti-proliferative effects on keratinocytes .

The exact mechanism of action of NBUVB is not known. It is proposed that it acts in the following ways: (1) Cellular DNA is converted to pyrimidine dimers which interfere with cell cycle progression, (2) alteration in cytokine production, NBUVB phototherapy as the second-line treatment for psoriasis, recommended when the topical therapy fails, is contraindicated or impractical. UVB radia- tions of wavelength 311 nm may result in the clearance of disease symptoms after just 5-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* : patients from 10 to 60 diagnosed to have psoriasis vulgaris

Exclusion Criteria:

1. concomitant chronic inflammatory disease or malignancy.
2. pregnant and lactating women.
3. renal dysfunction.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
measure serum vitamin D before and after treatment in psoriatic patients | 1 year
  A 3ml blood sample will be collected from the patients, then allowed to clot for 10 minutes and then centrifuged .
  Group 1: 20 patients under oral vitamin D therapy ( oral alpha one for 3 months o.25 microgram / day ) in combination with narrow band UVB settings (twice/week) Group 2 : 20 patients under narrow band UVB therapy only . c) We evaluate psoriatic patient by PASI score before and after treatment :
  ) measurment vitamin D level before and after treatment.

SECONDARY OUTCOMES:
We evaluate psoriatic patient by PASI score before and after treatment : | 1 year
  The body is divided into four sections (head (H) (10% of a person's skin); arms (A) (20%); trunk (T) (30%); legs (L) (40%)).
  Each of these areas is scored by itself, and then the four scores are combined into the final PASI. For each section, the percent of area of skin involved, is estimated and then transformed into a grade from 0 to 6:
  0.0% of involved area
  1.< 10% of involved area 2.10-29% of involved area 3.30-49% of involved area 4.50-69% of involved area 5.70-89% of involved area 6.90-100% of involved area